CLINICAL TRIAL: NCT05014490
Title: Randomized, Open-label, Single-dose, Two-sequence, Two-period, Crossover, Comparative, Oral Bioequivalence Study of Exib 120 mg Etoricoxib Film-coated Tablets (PrJSC "Pharmaceutical Firm "Darnitsa") and Arcoxia 120 mg Etoricoxib Film-coated Tablets (Merck Sharp&Dohme B.V.) in Healthy, Adult Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Test and Reference 120 mg Etoricoxib Film-coated Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Darnitsa Pharmaceutical Company (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ETR01-E
Record Dates: First submitted 2021-08-03; First posted 2021-08-20 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bioequivalence; Healthy Subjects
Keywords: bioequivalence; etoricoxib; healthy subjects; pharmacokinetics
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Intervention Model Description: Two-period, two-sequence, two-way crossover single dose study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exib (Test) (Experimental): A single oral dose of the test product Exib 120 mg etoricoxib film-coated tablets.
  Interventions: Drug: Exib 120 mg etoricoxib film-coated tablets
- Arcoxia® (Reference) (Active Comparator): A single oral dose of the reference product Arcoxia® 120 mg etoricoxib film-coated tablets.
  Interventions: Drug: Arcoxia® 120 mg etoricoxib film-coated tablets

INTERVENTIONS:
Drug: Exib 120 mg etoricoxib film-coated tablets — Oral, COX-2 highly selective, non-steroidal anti-inflammatory generic drug
  Arms: Exib (Test)
Drug: Arcoxia® 120 mg etoricoxib film-coated tablets — Oral, COX-2 highly selective, non-steroidal anti-inflammatory innovative drug
  Arms: Arcoxia® (Reference)

SUMMARY:
The present study is a comparative bioavailability study performed to assess bioequivalence between a Test medication (Exib 120 mg etoricoxib film-coated tablets manufactured by PrJSC "Pharmaceutical firm "Darnitsa" [Ukraine]) and a Reference medication (marketed medicinal product Arcoxia® 120 mg etoricoxib film-coated tablets, Marketing Authorisation Holder: UAB "Merck Sharp&Dohme", Lithuania) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian males.
2. Subjects aged between 18 and 55 years (inclusively) at the date of signing ICF which was defined as the beginning of the screening period.
3. Subjects with a BMI at screening within 18.5 to 30.0 kg/m2, inclusively.
4. Willingness to adhere to the protocol requirements and to provide written, personally signed, and dated ICF to participate in the study before the start of any study-related procedures.
5. Availability for the entire duration of the study.
6. Motivated subjects with absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee.
7. Satisfactory medical assessment at screening with no clinically relevant abnormalities as determined by medical history, physical examination, ECG, and clinical laboratory evaluation (haematology, biochemistry and urinalysis) that were reasonably likely to interfere with the subject's participation in or ability to complete the study as assessed by the Investigator.
8. Subjects were required to agree to abstain from xanthine-containing products (i.e. coffee, tea, cola, energy drinks, chocolate, etc.) from 48 hours prior to the first study drug administration until the end of confinement.
9. Subjects were required to agree to abstain from poppy seed-containing products from 48 hours prior to the first study drug administration until the end of confinement.
10. Subjects were required to agree to abstain from alcohol from 48 hours prior to the first study drug administration until the end of study.
11. Subjects were required to abstain and agree to continue to abstain from St John's Wort, vitamins and herbal remedies from 2 weeks prior to the first study drug administration until the end of confinement.
12. Subjects were required to abstain and agree to continue to abstain from beverages or food containing orange, grapefruit or pomelo from 2 weeks prior to the first study drug administration until the end of confinement.
13. Subjects had to agree to use medically acceptable methods of contraception during the study and for 30 days after the end of the study. Medically acceptable methods of contraception included using a condom with a female partner of childbearing potential who is using oral contraceptives, hormonal patch, implant or injection, intrauterine device, or diaphragm with spermicide. Complete abstinence alone could be used as a method of contraception.

Exclusion Criteria:

1. History of significant hypersensitivity to etoricoxib or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (such as angioedema) to any drug.
2. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
3. History of major surgery of the gastrointestinal tract except for appendectomy.
4. History of significant gastrointestinal, liver or kidney disease that might affect the drug BA.
5. Presence of significant cardiovascular, respiratory, genitourinary, musculoskeletal, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease.
6. Presence of respiratory infection symptoms (COVID-19 infection symptoms) like fever, dry cough, nasal congestion or sore throat.
7. Having COVID-19 infection or having been in contact to people with known COVID-19 infection in the last 14 days.
8. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes) within 6 months prior to Day 1 Period 1.
9. History of controlled or uncontrolled hypertension or clinically relevant Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and/or Heart Rate (HR) readings outside the normal ranges at screening (Day -3) or prior to drug administration on Day 1 Period 1. Normal ranges are defined below:

   * SBP: 90 to 140 mmHg
   * DBP: 60 to 90 mmHg
   * HR: 50 to 100 beats/min
10. Forehead body temperature readings outside the range of 35.5 to 37.4 ºC at screening (Day -5, -4, -3, -2, -1) or prior to the first drug administration.
11. Any planned surgery involving general, spinal or epidural anaesthesia from 3 months prior to Day 1 Period 1 to 7 days after last dosing.
12. Known presence of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption.
13. Any clinically significant illness within 30 days prior to Day 1 Period 1.
14. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and Human Immunodeficiency Virus (HIV) antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin and rifampicin) within 30 days prior to Day 1 Period 1.
15. Use of Over the Counter (OTC) medications within 7 days prior to Day 1 Period 1. It was specifically reminded that this included cold preparations, Acetylsalicylic Acid (ASA), natural products used for therapeutic benefits and antacid preparations.
16. Intake of any prescription medication within 30 days prior to Day 1 Period 1.
17. Maintenance therapy with any drug or significant history of drug dependency.
18. Alcohol abuse, i.e. regular use of more than 10 units per week (one unit of alcohol equals 250 mL of beer, 125 mL of wine or 25 mL of spirits), a history of alcoholism or recovered alcoholics.
19. Positive alcohol, drugs of abuse or cotinine results at screening (Day -1).
20. Positive result on Day -5 and/or Day -2 of screening on COVID-19 RT-PCR test.
21. History of drug abuse or use of illegal drugs: use of soft drugs (e.g. marihuana) within 6 months of screening or hard drugs (e.g. amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opioids) within 1 year of screening.
22. A positive Human Immunodeficiency Virus antibody (HIV-Ab) screen, Hepatitis B surface antigen (HBsAg) or Hepatitis C Virus (HCV) tests.
23. Use of an investigational product within 60 days prior to Day 1 Period 1 or active enrolment in another drug or vaccine clinical study.
24. Use of depot injectable solutions with a half-life of >1 week within 6 months prior to Day 1 Period 1.
25. Subjects previously randomised in this study.
26. An inability to follow a standardised diet and meal schedule or inability to fast, as required during the study.
27. Donation of blood (at least 100 mL) or plasma by plasmapheresis within 30 days prior to Day 1 Period 1.
28. Volunteers who reported difficulty swallowing tablets as a whole.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hakan Çetinsaya İyi Klinik Uygulama ve Arastirma Merkezi, IKUM (Center for GCP), Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exib (Test) First: Exib 120 mg etoricoxib film-coated tablets (test product) dosed in first period followed by Arcoxia 120 mg etoricoxib film-coated tablets (reference product) dosed in the second period.
- Arcoxia® (Reference) First: Arcoxia 120 mg etoricoxib film-coated tablets (reference product) dosed in first period followed by Exib 120 mg etoricoxib film-coated tablets (test product) dosed in the second period.
Period: First Intervention
Arm/Group | Exib (Test) First | Arcoxia® (Reference) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Exib (Test) First | Arcoxia® (Reference) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exib (Test) First | Arcoxia® (Reference) First | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The Cmax values are based on the etoricoxib plasma concentration.
Time Frame: Blood sampling for pharmacokinetic analysis covered up to 72 hours post-dose.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Exib): 120 mg Exib film-coated tablets test product dosed in either period.
- Reference (Arcoxia®): 120 mg Arcoxia® film-coated tablets reference product dosed in either period.
Arm/Group | Test (Exib) | Reference (Arcoxia®)
Number analyzed (Participants) | 28 | 28
ng/mL | 1948.656 (577.431) | 1916.300 (602.446)
Statistical Analysis 1: Comparison: Test (Exib) vs Reference (Arcoxia®); Test type: Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. The level of significance was set to the standard value of 5% (0.05) for all statistical tests; Ratio of the T/R geometric mean x 100 = 102.15, 90% CI 2-sided [94.54 to 110.37] — The ratio of geometric LSmeans with corresponding 90% CI calculated from the exponential of the difference between the test and reference products for the ln-transformed parameters should be within the acceptance interval of 80.00 - 125.00%

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t)
Description: The AUC0-t is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (t) and is based on the etoricoxib plasma concentration.
Time Frame: Blood sampling for pharmacokinetic analysis covered up to 72 hours post-dose.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Test (Exib) | Reference (Arcoxia®)
Number analyzed (Participants) | 28 | 28
h*ng/mL | 21967.848 (5570.437) | 22205.479 (6046.728)
Statistical Analysis 1: Comparison: Test (Exib) vs Reference (Arcoxia®); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.23, 90% CI 2-sided [96.97 to 101.54] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Information on AEs was continuously collected throughout the study from the screening until the follow up visit up to 23 days for each subject.
Description: Safety population included all dosed participants.
Arm/Group | Test (Exib) | Reference (Arcoxia®)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 3/28 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Exib) (N=28) | Reference (Arcoxia®) (N=28)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT05014490/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT05014490/SAP_001.pdf